CLINICAL TRIAL: NCT00643097
Title: A Complementary Trial of an Immunotherapy Vaccine Against Tumor-Specific EGFRvIII
Brief Title: Vaccine Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Acronym: ACTIVATe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Sampson (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, John Sampson, Professor of Neurology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004040; P50NS020023 (NIH); CDR0000589632 (Other: National Cancer Institute); DUMC-5421 (Registry Identifier: DUMC IRB); NCT00090597 (obsolete NCT alias)
Record Dates: First submitted 2008-03-25; First posted 2008-03-26 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Malignant Neoplasms of Brain
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — sargramostim; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (ACTIVATE) (Experimental): Patients first receive 3 initial vaccinations of an epidermal growth factor receptor variant III (EGRRvIII)-specific peptide (PEP-3) keyhole limpet hemocyanin (KLH) conjugate vaccine and sargramostim (GM-CSF), referred to as PEP-3 vaccine, every 2 weeks starting 4 weeks after the completion of radiation. Subsequent vaccinations were given once a month until clinical or radiographic evidence of progression or death.
  Interventions: Biological: PEP-3 vaccine; Biological: sargramostim; Drug: Temozolomide
- Arm II (ACT II STD) (Experimental): Patients first receive 3 initial vaccinations of an epidermal growth factor receptor variant III (EGRRvIII)- specific peptide (PEP-3) keyhole limpet hemocyanin (KLH) conjugate vaccine and sargramostim (GM-CSF), referred to as PEP-3 vaccine, biweekly starting within 6 weeks of completing radiation. Additional vaccinations were given until clinical or radiographic evidence of progression or death. Patients subsequently receive temozolomide at a targeted dose of 200 mg/m2 for the first 5 days of a 28 day cycle.
  Interventions: Biological: PEP-3 vaccine; Biological: sargramostim; Drug: Temozolomide
- Arm III (ACT II DI) (Experimental): Patients first receive 3 initial vaccinations of an epidermal growth factor receptor variant III (EGRRvIII)- specific peptide (PEP-3) keyhole limpet hemocyanin (KLH) conjugate vaccine and sargramostim (GM-CSF), referred to as PEP-3 vaccine, biweekly starting within 6 weeks of completing radiation. Additional vaccinations were given until clinical or radiographic evidence of progression or death. Patients subsequently receive temozolomide at a targeted dose of 100 mg/m2 for the first 21 days of a 28 day cycle.
  Interventions: Biological: PEP-3 vaccine; Biological: sargramostim; Drug: Temozolomide

INTERVENTIONS:
Biological: PEP-3 vaccine — Given intradermally
Biological: sargramostim — Given intradermally
Drug: Temozolomide — Standard of care chemotherapy
  Other Names: TMZ; Temodar

SUMMARY:
RATIONALE: Vaccines made from a peptide may help the body build an effective immune response to kill tumor cells. Colony-stimulating factors, such as GM-CSF, increase the number of white blood cells and platelets found in bone marrow or peripheral blood. Giving vaccine therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess humoral and cellular immune responses to adjuvant PEP-3-KLH conjugate vaccine in patients with newly diagnosed glioblastoma multiforme (GBM).
* To assess the clinical efficacy of the PEP-3-KLH conjugate vaccine, in terms of progression-free survival, in patients with newly diagnosed GBM.

Secondary

* To determine whether patients with GBM, who are known to be at least mildly immunosuppressed, can respond to standard and proven vaccine strategies.
* To assess for any potential toxicity to the PEP-3-KLH conjugate vaccine in patients with newly diagnosed GBM.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center.

At the time the study was initiated, standard of care temozolomide was not established, therefore, Arm I (ACTIVATE)was given without monthly cycles of temozolomide. At the point of interim analysis, monthly cycles of temozolomide had become standard of care. Arm II was then given the standard of care 5-day cycles of monthly temozolomide and during this time, dose-intensified temozolomide was in trials to compare with the 5-day temozolomide. Therefore, Arm III was initiated to determine the immunologic effects of 21-day monthly cycles of temozolomide with vaccine.

* Arm I (ACTIVATE): Patients receive PEP-3-KLH conjugate vaccine and sargramostim (GM-CSF) intradermally on days 1, 15, and 29 and then monthly in the absence of disease progression or unacceptable toxicity.
* Arm II (ACT II Standard (STD)): Patients first receive 3 initial vaccinations of an epidermal growth factor receptor variant III (EGRRvIII)- specific peptide (PEP-3) keyhole limpet hemocyanin (KLH) conjugate vaccine and sargramostim (GM-CSF) biweekly starting within 6 weeks of completing radiation. Additional vaccinations are given until clinical or radiographic evidence of progression or death. Patients subsequently receive temozolomide at a targeted dose of 200 mg/m2 for the first 5 days of a 28 day cycle.
* Arm III (ACT II Dose-intensified (DI)): Patients first receive 3 initial vaccinations of an epidermal growth factor receptor variant III (EGRRvIII)- specific peptide (PEP-3) keyhole limpet hemocyanin (KLH) conjugate vaccine and sargramostim (GM-CSF) biweekly starting within 6 weeks of completing radiation. Additional vaccinations are given until clinical or radiographic evidence of progression or death. Patients subsequently receive temozolomide at a targeted dose of 100 mg/m2 for the first 21 days of a 28 day cycle.

  * Patients undergo delayed-type hypersensitivity (DTH) skin testing* at baseline, after the third vaccination, and then monthly thereafter. Patients also undergo leukapheresis to obtain sufficient peripheral blood lymphocytes for immunologic monitoring at baseline, after the third vaccination, and then, if applicable, at the time of positive DTH response, disease progression, or after the sixth course of post-radiotherapy temozolomide. Methods used for immunologic monitoring include Enzyme-linked Immunospot(ELISPOT) assays, cytotoxicity assays, fluorescence activated cell sorting (FACS), and ELISA.

NOTE: *Patients with positive DTH skin testing, also undergo skin punch biopsies.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed glioblastoma multiforme
* Has undergone prior gross total resection (GTR) followed by conformal radiotherapy* with or without concurrent chemotherapy

  * GTR is defined as ≥ 95% volumetric resection of the contrast-enhancing component on the preoperative MRI
  * Residual radiographic contrast enhancement on post-resection CT scan or MRI must be ≤ 1 cm in maximal diameter in any two perpendicular axial planes
  * No evidence of disease progression after completion of radiotherapy* NOTE: *Patients may enroll in part 2 of the study within 2 weeks after surgery; these patients will receive radiotherapy with concurrent chemotherapy during the study
* EGFRvIII-positive tumor by immunohistochemistry, polymerase chain reaction, or related molecular techniques
* Karnofsky performance status 80-100%
* Curran group status I-IV
* Signed informed consent form

Exclusion Criteria:

* Absolute Neutrophil Count (ANC) < 1,000/mm³
* Platelet count < 50,000/mm³
* Prothrombin Time/Partial Thromboplastin Time (PT/PTT) > 1.5 times normal
* Positive hepatitis B (HB) surface antigen (HbsAg), antibody to hepatitis B surface antigen (anti-HBs), and antibody to hepatitis B core antigen (anti-HBc)
* Pregnant or nursing
* Positive pregnancy test
* Active infection requiring treatment
* Unexplained febrile illness (T max > 101.5 F)
* Inflammatory bowel disease, lupus erythematosus, rheumatoid arthritis, or other autoimmune disease
* Known immunosuppressive disease
* Known HIV infection
* Diffuse leptomeningeal disease
* Unstable or severe concurrent medical condition, such as severe heart and lung disease or active hepatitis
* Demonstrated allergy to temozolomide or inability to tolerate temozolomide for reasons other than lymphopenia
* Concurrent corticosteroids (except for nasal or inhaled steroids) at a dose above physiologic levels (> 2 mg of dexamethasone/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2012-01 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Vlahovic, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Result] Schmittling RJ, Archer GE, Mitchell DA, Heimberger A, Pegram C, Herndon JE 2nd, Friedman HS, Bigner DD, Sampson JH. Detection of humoral response in patients with glioblastoma receiving EGFRvIII-KLH vaccines. J Immunol Methods. 2008 Nov 30;339(1):74-81. doi: 10.1016/j.jim.2008.08.004. Epub 2008 Sep 4. PMID 18775433
- [Result] Sampson JH, Heimberger AB, Archer GE, Aldape KD, Friedman AH, Friedman HS, Gilbert MR, Herndon JE 2nd, McLendon RE, Mitchell DA, Reardon DA, Sawaya R, Schmittling RJ, Shi W, Vredenburgh JJ, Bigner DD. Immunologic escape after prolonged progression-free survival with epidermal growth factor receptor variant III peptide vaccination in patients with newly diagnosed glioblastoma. J Clin Oncol. 2010 Nov 1;28(31):4722-9. doi: 10.1200/JCO.2010.28.6963. Epub 2010 Oct 4. PMID 20921459
- [Result] Sampson JH, Aldape KD, Archer GE, Coan A, Desjardins A, Friedman AH, Friedman HS, Gilbert MR, Herndon JE, McLendon RE, Mitchell DA, Reardon DA, Sawaya R, Schmittling R, Shi W, Vredenburgh JJ, Bigner DD, Heimberger AB. Greater chemotherapy-induced lymphopenia enhances tumor-specific immune responses that eliminate EGFRvIII-expressing tumor cells in patients with glioblastoma. Neuro Oncol. 2011 Mar;13(3):324-33. doi: 10.1093/neuonc/noq157. Epub 2010 Dec 10. PMID 21149254

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (ACTIVATE): Patients first receive 3 initial vaccinations of an epidermal growth factor receptor variant III (EGRRvIII)- specific peptide (PEP-3) keyhole limpet hemocyanin (KLH) conjugate vaccine and sargramostim (GM-CSF) every 2 weeks starting 4 weeks after the completion of radiation. Subsequent vaccinations were given once a month until clinical or radiographic evidence of progression or death.
- Arm II (ACT II STD): Patients first receive 3 initial vaccinations of an epidermal growth factor receptor variant III (EGRRvIII)- specific peptide (PEP-3) keyhole limpet hemocyanin (KLH) conjugate vaccine and sargramostim (GM-CSF) biweekly starting within 6 weeks of completing radiation. Additional vaccinations were given until clinical or radiographic evidence of progression or death. Patients subsequently receive temozolomide at a targeted dose of 200 mg/m2 for the first 5 days of a 28 day cycle.
- Arm III (ACT II DI): Patients first receive 3 initial vaccinations of an epidermal growth factor receptor variant III (EGRRvIII)- specific peptide (PEP-3) keyhole limpet hemocyanin (KLH) conjugate vaccine and sargramostim (GM-CSF) biweekly starting within 6 weeks of completing radiation. Additional vaccinations were given until clinical or radiographic evidence of progression or death. Patients subsequently receive temozolomide at a targeted dose of 100 mg/m2 for the first 21 days of a 28 day cycle.
Period: Overall Study
Arm/Group | Arm I (ACTIVATE) | Arm II (ACT II STD) | Arm III (ACT II DI)
Started | 18 | 12 | 10
Completed | 18 | 12 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (ACTIVATE) | Arm II (ACT II STD) | Arm III (ACT II DI) | Total
Number analyzed (Participants) | 18 | 12 | 10 | 40
Age, Continuous [Median (Full Range); unit: years] | 52 [29 to 67] | 57 [41 to 83] | 59 [49 to 66] | 53 [29 to 83]
Gender [Count of Participants; unit: Participants]
  Female | 5 | 1 | 4 | 10
  Male | 13 | 11 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Humoral and Cellular Immune Response
Description: Number of patients that developed a delayed-type hypersensitivity (DTH) response at following vaccination. Any skin reaction in response to the intradermal injection of the antigen was measured and recorded. A positive skin test was defined as > 5 mm induration (swelling).
Time Frame: 26 months
Population: The test was performed on a subset of patients in each group that were available at vaccine 8, and results posted for those 30 patients who had the tests performed.
Measure: Number; unit: participants
Arm/Group | Arm I (ACTIVATE) | Arm II (ACT II STD) | Arm III (ACT II DI)
Number analyzed (Participants) | 17 | 5 | 8
participants | 3 | 0 | 7

2. Primary Outcome: Clinical Efficacy of Vaccination, in Terms of Progression-free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to Macdonald criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
  Macdonald criteria are standard criteria in neuro-oncology. Tumor assessment was made according to the adapted MacDonald criteria based on the combined evaluation of: 1) assessment of the MRI scan for measurable, evaluable, and new lesions (made by the independent external expert too), 2) overall assessment of neurological performance (made by the investigator), 3) concomitant steroid use (as reported by the investigator).
Time Frame: 58 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (ACTIVATE) | Arm II (ACT II STD) | Arm III (ACT II DI)
Number analyzed (Participants) | 18 | 12 | 10
months | 14.2 [9.9 to 17.6] | 12.1 [10.5 to 23.7] | 11.6 [8.1 to 12.7]

3. Secondary Outcome: Response to Vaccination
Description: The objective is to assess the duration of immunosuppressive cytokine secretion and to identify a receptive interval for active immunotherapy. Immunosuppression will determined by monitoring a panel of immunosuppressive serum/plasma cytokines longitudinally and by determining the response of each patient to Recombivax Hepatitis B (HB) vaccination. Response is defined as seropositive or seronegative to the Hepatitis B surface antigen.
Time Frame: 26 months
Population: This objective was not completed, as the test was not performed successfully.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Arm I (ACTIVATE) | Arm II (ACT II STD) | Arm III (ACT II DI)
Number analyzed (Participants) | 18 | 12 | 10
Months | NA (NA) — This objective was not completed, as the test was not performed successfully. | NA (NA) — This objective was not completed, as the test was not performed successfully. | NA (NA) — This objective was not completed, as the test was not performed successfully.

4. Secondary Outcome: Toxicity to PEP-3 Vaccine Immunization
Description: To assess for any potential toxicity to the PEP-3 vaccine immunization in patients with newly diagnosed glioblastoma, Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was used to tabulate any toxicities attributable to PEP-3. The number of patients with toxicity attributable to vaccine while on study are tabulated.
Time Frame: 26 months
Measure: Number; unit: participants
Arm/Group | Arm I (ACTIVATE) | Arm II (ACT II STD) | Arm III (ACT II DI)
Number analyzed (Participants) | 18 | 12 | 10
participants | 4 | 1 | 7

ADVERSE EVENTS:
Time Frame: 26 months
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov.
Arm/Group | Arm I (ACTIVATE) | Arm II (ACT II STD) | Arm III (ACT II DI)
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/12 | 3/10
Other Adverse Events (participants affected / at risk) | 17/18 | 12/12 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (ACTIVATE) (N=18) | Arm II (ACT II STD) (N=12) | Arm III (ACT II DI) (N=10)
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (ACTIVATE) (N=18) | Arm II (ACT II STD) (N=12) | Arm III (ACT II DI) (N=10)
Ear and labyrinth disorders - Other, specify: Ear Fullness - not infection (Ear and labyrinth disorders) | 0 | 0 | 1
Ear and labyrinth disorders - Other, specify: Left ear fluid (Ear and labyrinth disorders) | 1 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0
Eye disorders - Other, specify: Decreased Visual Acuity (Eye disorders) | 1 | 0 | 0
Eye disorders - Other, specify: Right Visual Field Cut (Eye disorders) | 1 | 0 | 0
Eye disorders - Other, specify: Visual Changes (Eye disorders) | 2 | 0 | 0
Flashing lights (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other, specify: Eating while Asleep - side effect of medication (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 6 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3
Chills (General disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 9 | 4 | 4
Fever (General disorders) | 2 | 1 | 1
Flu like symptoms (General disorders) | 0 | 0 | 4
Gait disturbance (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify: Drowsiness from medications (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 0
Immune system disorders - Other, specify: Redness on opposite side of vaccine injection site (Immune system disorders) | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 1 | 1
Bladder infection (Infections and infestations) | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 2 | 1 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, specify: Epidermoid cyst in Head (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify: Ringworm (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other, specify: Shingles (Infections and infestations) | 0 | 2 | 1
Lip infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 2 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 2 | 4
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Investigations - Other, specify: Vitamin D Deficiency (Investigations) | 0 | 1 | 0
Weight gain (Investigations) | 1 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 1
White blood cell decreased (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify: Left-sided Abdominal Contractions (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: Right Elbow Swelling/Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 0 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 5 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 2
Dysphasia (Nervous system disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 7 | 2 | 4
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 2 | 1
Nystagmus (Nervous system disorders) | 0 | 1 | 0
Olfactory nerve disorder (Nervous system disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 3 | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 3 | 3
Seizure (Nervous system disorders) | 4 | 1 | 1
Syncope (Nervous system disorders) | 3 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Confusion (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 4 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 2
Libido decreased (Psychiatric disorders) | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify: Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 5 | 3
Flushing (Vascular disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No